CLINICAL TRIAL: NCT04864652
Title: Safety and Dosing Study of the CHILLS Cryotherapy for the Treatment of Obstructive Sleep Apnea (OSA): ARCTIC-1
Brief Title: Safety and Dosing Study of the CHILLS Cryotherapy for the Treatment of OSA
Acronym: ARCTIC-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cryosa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10419
Record Dates: First submitted 2021-03-17; First posted 2021-04-29 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Experimental): CHILLS Procedure
  Interventions: Device: CHILLS Procedure

INTERVENTIONS:
Device: CHILLS Procedure — CHILLS Cryotherapy procedure

SUMMARY:
ARCTIC-1 is a safety and dosing study to evaluate procedure tolerability in patients with clinically diagnosed moderate or severe OSA.

DETAILED DESCRIPTION:
The study is a safety and dose titration study to determine the optimum dose of Cryosa CHILLS cryotherapy in patients with clinically diagnosed moderate or severe OSA.

Up to 70 subjects are planned to be enrolled and treated with the device at up to 3 clinical sites in Latin America. Subjects will be followed for 90 days with evaluation intervals at discharge, 7 days, 30 days and 90 days post-procedure. Subjects agreeing to long-term follow-up will complete visits every 6 months through 2 years post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25 - 65 years.
2. Diagnosed with moderate to severe OSA based on history and physical or have an established diagnosis of OSA (AHI ≥ 15 and ≤ 50) based on a prior sleep study.
3. BMI is between 28 kg/m2 and 40 kg/m2 at enrollment.
4. Negative result for COVID-19 polymerase chain reaction (RT-PCR) test and absence of clinical symptoms for COVID-19.

Exclusion Criteria:

1. Subjects with a high percentage of central apneas suggesting heart failure.
2. Contraindication to general anesthesia and MRI.
3. Metal braces, plate or pieces in the head or jaw that may interfere with MRI.
4. Craniofacial abnormality (e.g. retrognathia, micrognathia, etc.) thought to be the primary cause of OSA.
5. Obvious fixed upper airway obstructions (tumors, polyps, nasal obstruction) .
6. Tonsil size ≥ +3.
7. Previous surgery within 12 weeks of scheduled procedure performed on the soft tissue of the upper airway (e.g., uvula, soft palate or tonsils).
8. Oral cancer or non-healing oral wounds.
9. Presence of symptoms of influenza-like symptoms.
10. Contra-indicated for anesthesia or surgery.
11. History of surgery affecting the tongue (TORS, semi-glossectomy, RFBOT, MMA, HGNS).
12. History of radiation therapy to neck or upper respiratory tract
13. Surgical resection for cancer or congenital malformations in the larynx, tongue, or throat (with exception of tonsillectomy and/or adenoidectomy).
14. Clinical evidence of severe chronic obstructive or restrictive pulmonary disease (for example chronic bronchitis, emphysema, pulmonary fibrosis).
15. Active, severe pulmonary vascular disease (for example pulmonary arterial hypertension or pulmonary embolism).
16. Currently receiving treatment for severe cardiac valvular dysfunction, NYHA Class III or IV heart failure, unstable angina or recent (< 12 month) myocardial infarction or severe cardiac arrhythmias.
17. Subjects with bleeding event, known bleeding diathesis, impaired immunity for any reason, or heart attack or stroke within the last 12 months.
18. Clinical evidence of severe renal failure (Stage 4 or 5) undergoing dialysis or expected to institute dialysis within 12 months.
19. History or current clinical evidence of TIA or stroke or muscular dysfunction.
20. Taking medications that in the opinion of the consulting physician may alter consciousness, the pattern of respiration, or sleep architecture, such examples being benzodiazepines, opiates, neuroleptics, prescription stimulants, phenothiazine, or any form of chemical substance abuse.
21. History of dementia or active psychiatric disease that may impact study compliance.
22. Females who are pregnant or females of childbearing age with intention to become pregnant during the study period (≤ 3 months from treatment date).
23. Unable and/or unwilling to comply with study requirements or to provide written informed consent.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Procedure-Related Complications | 30 Days
  No serious procedure-related complications including death, loss of the airway requiring post-anesthesia care unit (PACU) re-intubation, persistent loss (more than 30 days) of tongue movement, or bleeding requiring surgical intervention or transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Marquito Caballero, MD, Principal Investigator — Sanatorio Americano; Stella Rowley, MD, Principal Investigator — San Fernando Specialized Center
Locations (2):
- Paitilla Medical Center, Panama City, Panama
- Sanatorio Americano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No